CLINICAL TRIAL: NCT01086722
Title: Pharmacokinetics in Morbid Obesity: Influence of Two Bariatric Surgery Techniques in Drugs Metabolism.
Brief Title: Pharmacokinetics in Morbid Obesity After Bariatric Surgery
Acronym: FAROBE/1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion IMIM (Other)
Collaborators: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FAROBE/1; 2009-013156-72 (EudraCT Number)
Record Dates: First submitted 2010-03-03; First posted 2010-03-15 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Morbid Obesity; Overweight
MeSH Terms: conditions — Obesity, Morbid; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- "karolinska cocktail" (Experimental): The karolinska cocktail contains dextromethorphan, caffeine, losartan and omeprazol
  Interventions: Drug: "karolinska cocktail"

INTERVENTIONS:
Drug: "karolinska cocktail" — The "karolinska cocktail" contains dextrometorphan, caffeine, losartan and omeprazol

SUMMARY:
Morbid obesity (MO) is associated with several disorders such as hypertension, type 2 diabetes, dyslipemia and degenerative arthropathy that require pharmacological treatment. Drug bioavailability and metabolism in patients with MO is altered compared to population controls. Bariatric surgery is the gold standard treatment for MO when conventional therapy fails.

Bariatric surgery techniques can modify drug absorption in MO patients. These modifications depend on the drug absorption characteristics and on the bariatric surgery technique used. The changes in weight and body composition caused by BS at middle term can alter drug bioavailability and metabolism. The kinetics of the "normalization" process in patients with MO after bariatric surgery is unknown

Objectives. To analyze the changes in drug metabolism and pharmacokinetics. To establish drug dosing criteria in the post-intervention period in patients with MO after bariatric surgery. To determine the relationship between changes in drug bioavailability and metabolism in MO after bariatric surgery (longitudinal gastrectomy and Y-roux gastric by-pass).

DETAILED DESCRIPTION:
Patients and methods. A prospective study of two cohorts of patients in a program of bariatric surgery (gastric by-pass and sleeve gastrectomy). Study "before and after".

Evaluations. Study on drug metabolism and pharmacokinetics using a modified "karolinska cocktail" (dextromethorphan, caffeine, losartan, omeprazole and paracetamol) before bariatric surgery and at 4 weeks and 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults (from 18 to 55 years)
* Morbid Obesity BMI > 40 or BMI> 35 plus co-morbidity
* Healthy controls (non-overweight and overweight groups)

Exclusion Criteria:

* Allergy to study drugs
* Liver diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Metabolic ratios of probe substances | 8 hours after drug administration
  Metabolic ratios of parent drugs and metabolites in plasma and urine before and after bariatric surgery.

SECONDARY OUTCOMES:
Pharmacokinetics of probe substances | 0-8 hours
  Comparison of the pharmacokinetics. Comparison of the metabolic ratios of probe substances between obese morbid patients and controls (normal weight and overweight).
  Adverse events observed after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Albert Goday, MD, Principal Investigator — Hospital del Mar
Locations (2):
- Spain (2):
  - Hospital del Mar, Barcelona, Barcelona
  - IMIM-Hospital del Mar, Barcelona, Barcelona

REFERENCES:
- [Derived] Goday Arno A, Farre M, Rodriguez-Morato J, Ramon JM, Perez-Mana C, Papaseit E, Civit E, Langohr K, Li Carbo M, Boix DB, Nino OC, Le Roux JAF, Pera M, Grande L, de la Torre R. Pharmacokinetics in Morbid Obesity: Influence of Two Bariatric Surgery Techniques on Paracetamol and Caffeine Metabolism. Obes Surg. 2017 Dec;27(12):3194-3201. doi: 10.1007/s11695-017-2745-z. PMID 28560524